CLINICAL TRIAL: NCT03907462
Title: SMART 2.0: Social Mobile Approaches to Reducing weighT in Young Adults
Acronym: SMART 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Small Steps Labs, LLC (Unknown)
Responsible Party: Principal Investigator, Job Godino, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 181862; 1R01HL136769-01A1 (NIH)
Record Dates: First submitted 2019-03-27; First posted 2019-04-09 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity
Keywords: young adult; overweight; obesity; college; university; technology; social media; text message; health coach; intervention; weight loss; wellness; physical activity; diet; sleep; resilience; wearable; mobile application; behavior mechanism; behavior
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Motor Activity; Behavior

STUDY DESIGN:
Intervention Model Description: The study is a 24-month parallel-group randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment One (Experimental): Participants assigned to the SMART 2.0 with technology and personal health coaching treatment group (i.e., treatment one) will receive the following: 1) consumer-level wearable and scale with a corresponding app, 2) daily text messages related to physical activity, diet, sleep and weight loss/maintenance, 3) access to SMART 2.0 social media pages and content through an online group with 6 to 12 participants total, and 4) technology-mediated, real-time individual health coaching. Participants will receive 1 to 2 text messages on a daily basis; be asked to use their wearable on a daily basis and self-weigh using the scale at least once per week; be asked to interact with their online group via social media as frequently as possible; and speak with their health coach at a predetermined session schedule.
  Interventions: Behavioral: SMART 2.0
- Treatment Two (Experimental): Participants assigned to the SMART 2.0 technology alone treatment group (i.e., treatment two) will receive the following: 1) consumer-level wearable and scale with a corresponding app, 2) daily text messages related to physical activity, diet, sleep and weight loss/maintenance, and 3) access to SMART 2.0 social media pages and content through an online group with 6 to 12 participants total. Participants will receive 1 to 2 text messages on a daily basis; be asked to use their wearable on a daily basis and self-weigh using the scale at least once per week; and be asked to interact with their online group via social media as frequently as possible.
  Interventions: Behavioral: SMART 2.0
- Control (No Intervention): Participants assigned to the control group will receive a consumer-level wearable and scale with a corresponding app to use at their discretion.

INTERVENTIONS:
Behavioral: SMART 2.0 — SMART 2.0 uses a fully integrated system of modalities that includes: 1) a popular consumer-level wearable, wireless scale, and corresponding app; 2) a highly tailored and interactive text messaging system; 3) multiple social media streams; 4) social network mechanisms of influence; and 5) technology-mediated health coaching.
  Arms: Treatment One; Treatment Two

SUMMARY:
The SMART 2.0 study is a 24-month trial designed to evaluate the impact of the intervention with technology and personal health coaching or with technology alone on objectively measured weight among overweight young adults in a university setting over 24 months compared to a control group. The investigators hypothesize that both interventions will significantly improve weight compared to the control group, and the group receiving personal health coaching will experience the greatest improvement.

DETAILED DESCRIPTION:
Weight gain is an important issue for young adults. Throughout the transition from adolescence to early adulthood, young adults encounter multiple stressors and influences that can contribute to weight gain. In turn, weight gain leads to increased risk of cardiovascular disease, diabetes, and other health issues. Thus, there is a critical need to advance our understanding of how to develop and deploy multimodal, technology-based weight-loss interventions that have the potential for long-term effects and widespread dissemination among young adults.

The SMART 2.0 study is a 24-month (96 week) parallel-group randomized control trial designed to evaluate the impact of the interventions on objectively measured weight in kg over 24 months compared to a control group. The study will recruit 642 overweight/obese young adults aged 18-35 at universities in San Diego, CA. Participants will be randomly assigned to one of three groups for a 24-month study period. The three groups include: 1) SMART 2.0 with a consumer-level wearable and scale, text messaging, social media, and technology-based health coaching; 2) SMART 2.0 with a consumer-level wearable and scale, text messaging, and social media; and 3) a control group with a consumer-level wearable and scale alone. Theory- and evidence-based content will be framed around a minimum goal of 5-10% weight loss through increased energy expenditure, decreased energy intake, and adequate sleep. Additionally, participants will be encouraged to lose 1 to 2 pounds per week until they reach a body mass index (BMI) below 25 kg/m2. Once a participant reaches a BMI less than 25 kg/m2 the goal will be to maintain their weight loss.

SMART 2.0 uses a fully integrated system of modalities that includes: 1) a popular consumer-level wearable (e.g., Fitbit Charge 3), wireless scale (e.g., Aria Scale), and corresponding app (e.g., the Fitbit app); 2) a highly tailored and interactive text messaging system; 3) multiple social media streams (e.g., Facebook, Facebook Messenger, Instagram, and Twitter); and 4) social network mechanisms of influence. The consumer-level devices and app will be used to self-monitor behavior, and their data will be passively acquired in real-time. Algorithms will be used to automatically deliver text messages to support individually tailored goal setting, performance feedback, and goal review in a highly dynamic style that reflects participants' behavioral progress towards achieving a minimum goal of 5% weight loss. Participants will be encouraged to share their data and behavioral progress with others via social networking tools. Social network mechanisms of influence will be used both within the study-space, to elicit participant-to-participant and health coach-to-participant support, as well as outside the study-space, to invoke social support and accountability from strong ties known to be important for long-term behavior change. Additionally, one group will receive monthly technology-mediated and real-time personal health coaching that is theory- and evidence-based.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35 years
* Intending to be available for a 24 month intervention
* Affiliated with either University of California, San Diego (UCSD), San Diego State University (SDSU), or California State University, San Marcos (CSUSM) as a student, faculty, or staff
* Willing and able to use social media
* Willing and able to use a smartphone and text messaging
* Willing and able to use the wearable, scale, and corresponding app
* Willing and able to attend measurement visits over the 2 year intervention
* Willing and able to engage in moderate to vigorous physical activity
* Overweight or obese, but not severely obese (25 >= BMI < 40 kg/m2)

Exclusion Criteria:

* Any comorbidities of obesity that require a clinical referral including eating disorders, pseudotumor cerebri, sleep apnea or hypoventilation syndrome, orthopedic problems, and meeting American Diabetes Association criteria for diabetes
* Psychiatric or medical conditions that prohibit compliance with the study protocol
* Had a cardiovascular event (heart attack, stroke, episode of heart failure, or revascularization procedure) within the last 6 months
* Currently being treated for a malignancy (other than non-melanoma skin cancer)
* Currently being treated and/or have an eating disorder
* Planning to have a weight loss surgery in the next 24 months (e.g., liposuction, lap band, gastric bypass)
* Pregnant, gave birth within the last 6 months, currently lactating or breastfeeding within the last 3 months, or actively planning pregnancy within the next 24 months
* Prescribed physical activity and/or dietary changes
* Prescribed medications that alter weight
* Enrolled in or planning to enroll in a weight loss program during the study period
* Lost more than 15 pounds within the past 3 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 638 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Job G Godino, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godino JG, Merchant G, Norman GJ, Donohue MC, Marshall SJ, Fowler JH, Calfas KJ, Huang JS, Rock CL, Griswold WG, Gupta A, Raab F, Fogg BJ, Robinson TN, Patrick K. Using social and mobile tools for weight loss in overweight and obese young adults (Project SMART): a 2 year, parallel-group, randomised, controlled trial. Lancet Diabetes Endocrinol. 2016 Sep;4(9):747-755. doi: 10.1016/S2213-8587(16)30105-X. Epub 2016 Jul 14. PMID 27426247
- [Derived] Baretta D, Chevance G, Mansour-Assi SJ, Costello VL, Wing D, Hekler EB, Inauen J, Godino J, Nigg CR. Exploring boundary conditions of physical activity maintenance: A secondary analysis of time-series data from a weight-loss intervention. Health Psychol Behav Med. 2025 Sep 11;13(1):2554980. doi: 10.1080/21642850.2025.2554980. eCollection 2025. PMID 40948958
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Mansour-Assi SJ, Golaszewski NM, Costello VL, Wing D, Persinger H, Coleman A, Lytle L, Larsen BA, Jain S, Weibel N, Rock CL, Patrick K, Hekler E, Godino JG. Social Mobile Approaches to Reducing Weight (SMART) 2.0: protocol of a randomized controlled trial among young adults in university settings. Trials. 2022 Jan 3;23(1):7. doi: 10.1186/s13063-021-05938-7. PMID 34980208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Young adults aged 18-35 years were recruited from 3 universities and 5 community colleges in San Diego, CA through digital advertisements, print and digital flyers, email listservs, and campus-wide events. Interested individuals were directed to secure online screening form. Eligibility criteria were confirmed through telephone screening with study staff. Eligible were invited to schedule a baseline appointment. There participants were rescreened, provided written informed consent, and enrolled.
Pre-assignment Details: After eligibility and consent were confirmed and baseline measurements were completed, participants were stratified by sex and university/college and then randomized within each stratum at a ratio of 1:1:1 to one of three study arms.
Period: Overall Study
Arm/Group | Treatment One | Treatment Two | Control
Started | 214 | 212 | 212
Completed | 187 | 186 | 180
Not Completed | 27 | 26 | 32
Not completed — Physician Decision | 1 | 3 | 1
Not completed — Withdrawal by Subject | 6 | 3 | 3
Not completed — Pregnancy | 4 | 2 | 6
Not completed — Lost to Follow-up | 16 | 18 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment One | Treatment Two | Control | Total
Number analyzed (Participants) | 214 | 212 | 212 | 638
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.285 (4.539) | 22.439 (4.208) | 23.099 (4.628) | 22.942 (4.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 126 | 126 | 378
  Male | 88 | 86 | 86 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 86 | 80 | 96 | 262
  Not Hispanic or Latino | 128 | 132 | 116 | 376
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 60 | 50 | 53 | 163
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 6 | 7 | 5 | 18
  White | 44 | 49 | 48 | 141
  More than one race | 101 | 99 | 103 | 303
  Unknown or Not Reported | 2 | 5 | 3 | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) calculated as kg/m^2
  kg/m^2 | 30.329 (3.71) | 30.273 (3.624) | 30.283 (3.772) | 30.295 (3.696)
Weight [Mean (Standard Deviation); unit: Kilograms] — Measured in kilograms.
  Kilograms | 86.393 (13.034) | 85.008 (13.304) | 84.925 (14.135) | 85.445 (13.494)
Waist circumference [Mean (Standard Deviation); unit: Centimeters] — Measured following standardized procedures from the approximate midpoint between the low margin of the last palpable rib and the top of the iliac crest.
  Centimeters | 83.264 (6.307) | 83.235 (8.257) | 83.350 (6.393) | 83.283 (7.03)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Objectively measured weight in kilograms.
Time Frame: Baseline, 24 months
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Treatment One | Treatment Two | Control
Number analyzed (Participants) | 187 | 186 | 180
Kilograms | -0.333 (6.553) | 0.737 (7.631) | 1.202 (8.045)

2. Secondary Outcome: Change in Body Mass Index
Description: Weight and height will be combined to report BMI in kg/m^2.
Time Frame: Baseline, 24 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Treatment One | Treatment Two | Control
Number analyzed (Participants) | 129 | 125 | 125
kg/m^2 | -0.213 (2.199) | 0.015 (2.607) | 0.418 (2.548)

3. Secondary Outcome: Percent Weight Change
Description: Percent change in weight from baseline.
Time Frame: Baseline, 24 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment One | Treatment Two | Control
Number analyzed (Participants) | 153 | 153 | 144
percent change | -0.265 (7.414) | 0.955 (8.674) | 1.437 (8.829)

4. Secondary Outcome: Percentage of Participants Who Lost at Least 3% of Their Weight From Baseline
Description: Percentage of participants who lost at least 3% of their weight from baseline.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Percentage of Participants Who Lost at Least 5% of Their Weight From Baseline
Description: Percentage of participants who lost at least 5% of their weight from baseline.
Time Frame: Baseline, 24 months
Population: Only participants with a 24 month primary outcome measure are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment One | Treatment Two | Control
Number analyzed (Participants) | 153 | 153 | 144
Participants | 35 | 28 | 27

6. Secondary Outcome: Change in Waist Circumference
Description: Objectively measured in centimeters.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: Change in Waist-to-hip Ratio
Description: Waist and hip circumference will be combined to report waist-to-hip ratio in cm/cm.
Time Frame: Baseline, 24 months
Population: Only participants with a 24 month waist and hip outcome measures are included in this analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment One | Treatment Two | Control
Number analyzed (Participants) | 145 | 140 | 139
Ratio | -0.622 (4.033) | -0.064 (2.789) | 0.141 (2.643)

8. Secondary Outcome: Change in Body Composition
Description: Total body and regional (arms, legs, trunk, and abdomen) body composition (fat mass, including an estimate of visceral adipose tissue, and lean mass) measured with Dual-energy X-ray Absorptiometry (DXA).
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Change in Bone Mineral Density
Description: Bone mineral density of anterior-posterior spine (L1 - L4), hip, forearm, and total body measured with Dual-energy X-ray Absorptiometry (DXA).
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure in mmHg.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

11. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Diastolic blood pressure in mmHg.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

12. Secondary Outcome: Change in Cardiorespiratory Fitness
Description: Three-minute step test.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

13. Secondary Outcome: Change in Flexibility
Description: Sit and reach test.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

14. Secondary Outcome: Change in Grip Strength
Description: Grip strength of the right and left hands in kilograms with a dynamometer.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

15. Secondary Outcome: Physical Activity
Description: Measured using Fitbit.
Time Frame: Through study completion, up to 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

16. Secondary Outcome: Physical Activity
Description: Measured using a waist-worn tri-axial accelerometer.
Time Frame: For 7 days, at 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

17. Secondary Outcome: Change in Physical Activity
Description: Assessed through self-report using the Global Physical Activity Questionnaire. The questionnaire is comprised of 16 questions related to physical activity in three settings that include activity at work, travel to and from places, and recreational activities, in addition to sedentary behavior. Metabolic Equivalent (MET) values are assigned to time variables according to intensity of activity, moderate or vigorous, reported in each of the settings. MET values are then used to calculate total physical activity.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

18. Secondary Outcome: Sleep
Description: Measured using Fitbit.
Time Frame: Through study completion, up to 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

19. Secondary Outcome: Change in Sleep
Description: Assessed through self-report using an 8 item self-report questionnaire. Participants respond to questions related to sleep duration and how often they have difficulty falling asleep and staying awake, do not get enough rest.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

20. Secondary Outcome: Resting Heart Rate
Description: Measured using Fitbit.
Time Frame: Through study completion, up to 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

21. Secondary Outcome: Change in Resting Heart Rate
Description: Measured by research assistant.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

22. Secondary Outcome: Sedentary Behavior
Description: Measured using Fitbit.
Time Frame: Through study completion, up to 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

23. Secondary Outcome: Sedentary Behavior
Description: Measured using a waist-worn tri-axial accelerometer.
Time Frame: For 7 days, at 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

24. Secondary Outcome: Change in Sedentary Behavior
Description: Assessed through self-report using 5 items from the Canadian Fitness Survey and 10 items from the Past-day Adults' Sedentary Time Questionnaire. Participants respond to items from the Canadian Fitness Survey related to how much time participants spend doing sedentary activities on a 5-point response scale ranging from "Almost all of the time" to "Almost none of the time". Participants respond to items from the Past-day Adults' Sedentary Time Questionnaire related to how much time spent sitting while doing activities including working, transportation, etc. using 2 digit entry for hours and minutes. For all items, less time reported doing sedentary activities or sitting represents less sedentary behavior.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

25. Secondary Outcome: Diet History Questionnaire III
Description: The Diet History Questionnaire III contains 135 food and beverage items and 26 dietary supplement items to assess diet consumption for past month. The questionnaire includes additional embedded questions for some items to assess frequency and portion size.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

26. Secondary Outcome: Weight Management Practices
Description: Assessed through self-report using a 3-item questionnaire. Participants respond to items related to which behaviors they have engaged in in the past 30 days to lose weight, how often they weigh themselves using a 6 point response scale ranging from "Never" to "More than once a day", and whether they have access to a scale at home.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

27. Secondary Outcome: Strategies for Weight Management Questionnaire
Description: Strategies for Weight Management Questionnaire consists of 35 items that assess how often participants use of behavioral strategies for reducing energy intake and increasing energy expenditure on a 5-point response scale ranging from "Never or hardly ever" to "Always or almost always". Values which indicate a higher frequency of strategies, "Much of the time" and "Always or almost always", show improved weight management.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

28. Secondary Outcome: Assessment of Eating Behaviors
Description: Assessment of Eating Behaviors survey consists of 8 items that assess sugar sweetened beverage consumption and frequency of eating away from home on a 9-point response scale ranging from "Never or rarely" to "3 or more times per day".
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

29. Secondary Outcome: Daily Meal Patterns
Description: Assessed through self-report using a 7-item questionnaire. Participants respond to items related to how often they eat meals and snacks in a typical week using a 5-point response scale ranging from "0 times" to "7 times".
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

30. Secondary Outcome: Healthy Eating: Change Strategies
Description: Healthy Eating: Change Strategies survey consists of 15-items that assess how often participants engage in strategies that help them change their dietary habits in the past month using a 5-point response scale ranging from "Never" to "Many times".
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

31. Secondary Outcome: Physical Activity: Change Strategies
Description: Physical Activity: Change Strategies survey consists of 15-items that assess how often participants engage in strategies that help them change their physical activity in the past month using a 5-point response scale ranging from "Never" to "Many times".
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

32. Secondary Outcome: Physical Activity Neighborhood Environment
Description: Physical Activity Neighborhood Environment survey consists of 17-items that assess the environmental factors for walking and bicycling in various neighborhoods. Higher values from the scale indicate greater environmental support for physical activity.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

33. Secondary Outcome: Social Support for Healthy Eating Habits
Description: Social Support for Diet survey consists of 10-items that assess perceived social support specific to health-related eating behaviors from family and friends, respectively. Each item uses a 8-point response scale that includes "does not apply" and ranges from "none" to "very often".
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

34. Secondary Outcome: Social Support for Physical Activity
Description: Assessed using the Physical Activity and Social Support Scale which consists of 20-items scale based in five forms of social support - companionship, emotional, instrumental, informational, and validation for physical activity. Participants respond to items on a 7-point Likert scale ranging from "never" to "always", or "not applicable".
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

35. Secondary Outcome: Depression
Description: Assessed using the Center for Epidemiologic Studies depression scale which consists of 10-items. Participants respond to items related to how they feel and behave on a 5-point response scale ranging from "Rarely or none of the time" to "All of the time". A score equal to or above 10 is considered depressed.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

36. Secondary Outcome: Anxiety
Description: Assessed using the short-form of the state scale of the Spielberger State Trait Anxiety Inventory which consists of 6 items. Participants respond to items related to how they feel on a 4-point response scale ranging from "Not at all" to "Very much".
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

37. Secondary Outcome: Self-esteem
Description: Assessed using the Rosenberg Self-esteem Scale which consists of 10-items. Participants respond to items related to items related to global self-worth on a 4-point Likert scale ranging from "strongly agree" to "strongly disagree". Higher scores indicate higher self-esteem.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

38. Secondary Outcome: Quality of Well-being
Description: Assessed using the Quality of Well-being survey, self-administered version which consists of 71 items. Participants respond to items related to health status and overall well-being over the previous 3 days. Scores are translated to quality-adjusted life years.
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

39. Secondary Outcome: Body Image
Description: Assessed using the Eating Disorder Inventory, Body Dissatisfaction sub scale which consists of 9-items. Participants respond to items related to their body image on a 6-point response scale ranging from "Never" to "Always".
Time Frame: Baseline, 24 months
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: The duration of the study (24 months).
Description: Adverse event was collected at each follow-up timepoint for all participants and via participant self-report throughout the trial period.
Arm/Group | Treatment One | Treatment Two | Control
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/212 | 0/212
Serious Adverse Events (participants affected / at risk) | 2/214 | 4/212 | 2/212
Other Adverse Events (participants affected / at risk) | 73/214 | 53/212 | 40/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment One (N=214) | Treatment Two (N=212) | Control (N=212)
Serious mental health episode (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) — New diagnosis for mental health disorder after displaying life-threatening behaviors.
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Participant experience non-related stroke
Muscle/bone injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Appendectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Serious COVID-19 case
Drug overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Overdose on fentanyl
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment One (N=214) | Treatment Two (N=212) | Control (N=212)
Muscle or bone injury (Musculoskeletal and connective tissue disorders) | 35 (38) | 23 (25) | 8 (11)
New diagnosis for mental health problem (Psychiatric disorders) | 8 (9) | 10 (11) | 7 (8)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 2 (2) | 6 (6)
Fainting (Social circumstances) | 1 (1) | 3 (3) | 0 (0)
New diagnosis of eating disorder (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
New diagnosis for diabetes (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 0 (0) | 4 (4)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) — Due to wearing Fitbit device for intervention
Migraine (General disorders) | 0 (0) | 2 (2) | 2 (2)
Weight loss treatment (Surgical and medical procedures) | 2 (2) | 0 (0) | 1 (1)
Asthmatic Episode (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Outpatient surgery (Surgical and medical procedures) | 3 (3) | 4 (4) | 1 (1) — Not weight loss related
New skin condition (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) — Not related to Fitbit
New metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Non-muscular Injury (General disorders) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03907462/Prot_SAP_000.pdf